CLINICAL TRIAL: NCT00760305
Title: Pro-self - a Nursing Intervention to Support and Educate Cancer Patients and Their Caregivers so That the Patient Can Stay Home
Brief Title: Pro-self Pain Management in Norway
Acronym: Pro-self
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Tone Rustøen professor, Oslo University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 158707/V10
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2008-09

CONDITIONS: Cancer; Pain
Keywords: cancer pain; bone metastasis; patient education; psychoeducational education; side effects; analgesics
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients who received the Pro-Self psychoeducational intervention
  Interventions: Behavioral: Pro self pain control programme
- 2 (No Intervention): Patients who received standard care

INTERVENTIONS:
Behavioral: Pro self pain control programme — A 6 week psychoeducational programme that included three home visits and three phone calls. Patients were taught about pain medication and side effects and about incorrect information regarding cancer pain management
  Arms: 1

SUMMARY:
The main aim of this study is to evaluate whether a patient education programme on cancer pain management compared to standard care decreases pain and increases patients quality of life. The investigators hypothesis is that patients and family caregivers who receive the intervention will have improved outcomes. Patients and family members are seen in their homes by the nurses doing the intervention over 6 weeks. Patients keep a diary of their pain and medication intake.

DETAILED DESCRIPTION:
The undertreatment of cancer pain remains a significant clinical problem. The PRO-SELF Pain Control Program is a 6 week psychoeducational intervention that was shown to improve pain management in oncology outpatients with pain from bone metastasis. However, this promising intervention requires replication in samples of oncology patients with cancer pain outside of the United States.

The purpose of the study was to test the effectiveness of The PRO-SELF Pain Control Program in Norwegian cancer patients and their family caregivers. Only data on patient outcomes will be presented.

The theoretical framework for this study incorporated elements of Orem's self-care theory, as well as the principles of academic detailing and nurse coaching to change patients' self-care behaviors regarding cancer pain management.

Two hundred adult cancer patients with pain from skeletal metastasis and their caregivers participated in this study. Patients were randomized to either the PRO-SELF program or standard care. Patients completed questionnaires about pain, physical functioning, quality of life, anxiety, and depression at the time of enrollment and after 6 weeks. Data on analgesics were collected through chart reviews and patient diaries. Both groups received home visits and telephone calls by an oncology nurse over a period of six weeks. Participants in the intervention group received education about pain management and were coached to improve their pain management behaviors. Two-way repeated measures analyses of variance will be done to determine differences in pain intensity scores and to evaluate the differences over time in the total amount of opioid analgesics taken by the patients.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Radiographic evidence of bone metastasis
* Able to read and write Norwegian
* Average pain intensity of greater than 2.5

Exclusion Criteria:

* Brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Worst pain intensity | 6 weeks

SECONDARY OUTCOMES:
Knowledge of cancer pain management | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tone Rustoen, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Ulleval University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Rustoen T, Lerdal A, Gay C, Kottorp A. Rasch analysis of the Herth Hope Index in cancer patients. Health Qual Life Outcomes. 2018 Oct 3;16(1):196. doi: 10.1186/s12955-018-1025-5. PMID 30285767